CLINICAL TRIAL: NCT00690183
Title: Relationship Between Physical Activity and Stem Cells in Older Adults
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0226-08-EP
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Aging
Keywords: physical activity; stem cells; lifestyle
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma will be retained for cytokine analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot study to develop a collaborative, translational research project investigating whether physical activity may in part exert a positive influence on aging via the mobilization of stem cells. Preliminary data will be collected to explore the relationship between physical activity and stem cell populations found in the blood. The study hypothesis is that stem cell decrease with age, but that persons who are more physically active will have a higher number of stem cells in the blood. The first assessment will include an evaluation of health, physical activity and lifestyle via questionnaires. Height, weight and abdominal girth will be measured, and blood will be drawn for immune and stem cell assessment. Participants will be given a pedometer and accelerometer to wear daily for 7 days. Participants will return for a second visit at which the pedometer and accelerometer will be returned and blood will be drawn. Stem cell and immune assays will be repeated to evaluate the variability of these measures over time. The correlation between stem cell numbers and physical activity will be analyzed.

DETAILED DESCRIPTION:
Increased numbers of circulating stem cells and physical activity are both associated with improved health in older persons. This pilot study is the initial step in developing a collaborative, translational research project investigating whether physical activity may in part exert a positive influence on aging via the mobilization of stem cells. The specific aim of this pilot project is to collect preliminary data to explore the relationship between physical activity and stem cell populations found in the blood and to determine the variance in the number of circulating stem cells. We hypothesize that stem cell decrease with age, but that persons who are more physically active will have a higher number of stem cells in the blood. A maximum of 40 persons will be recruited to participate. Persons are eligible to participate if they are age 60 or older, haven't been hospitalized recently, do not have an immunologic or blood disease, do not have an infection, and are not undergoing chemotherapy. Subjects will have 2 visits to the UNMC Clinical Research Center (CRC). The first assessment will include an evaluation of health, physical activity and lifestyle via questionnaires. Height, weight and abdominal girth will be measured, and blood will be drawn for immune and stem cell assessment. Subjects will be given a pedometer and accelerometer to wear daily for 7 days. Subjects will return to the CRC for a second visit at which the pedometer and accelerometer will be returned and blood will be drawn. Stem cell and immune assays will be repeated to evaluate the variability of these measures over time. The correlation between stem cell numbers and physical activity will be analyzed. The data will be used to perform sample size calculations for the development of future studies.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older

Exclusion Criteria:

* Hospitalization within 2 months prior
* Immunological disease
* Hematopoietic disease
* No current infection
* No current chemotherapy

Ages: 60 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample of Omaha, NE metro area
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2008-06-05 (Actual); Primary Completion 2008-08-01 (Actual); Study Completion 2008-10-01 (Actual)

PRIMARY OUTCOMES:
circulating stem cells | upon enrollment, one week later
  Number of circulating stem cells determined by lab
physical activity | upon enrollment
  physical activity as reported

SECONDARY OUTCOMES:
alcohol consumption | upon enrollment
  alcohol consumption as reported
smoking history | upon enrollment
  smoking history as reported
plasma cytokine levels | upon enrollment, one later
  plasma cytokine levels determined by lab

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Bilek, PhD, PT, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States